CLINICAL TRIAL: NCT05433558
Title: Effectiveness of Neuropsychological Rehabilitation Program for Disease of Adaptation in Patients With Acquired Brain Injury and Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-ER-110-145
Record Dates: First submitted 2022-06-14; First posted 2022-06-27 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-08

CONDITIONS: Acquired Brain Injury; Neuropsychological Rehabilitation; Caregiver
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): enter the experiment directly
  Interventions: Other: Neuropsychological Rehabilitation
- Waiting group (Experimental): enter the experiment after waiting eight weeks
  Interventions: Other: Neuropsychological Rehabilitation

INTERVENTIONS:
Other: Neuropsychological Rehabilitation — Neuropsychological Rehabilitation

SUMMARY:
Acquired brain injury is mental function damage caused by different reasons (such as cerebral neuropathy, head injury, traumatic brain injury, stroke, brain tumor, etc.). After the injury, patient has mental, cognitive, behavioral, body function, and other impairments, which makes patient still need the assistance of family members. For patients with brain injury in subacute stage, clinician assesses their needs for follow-up rehabilitation intervention programs in an appropriate way to assist patients who have the potential to return home to make care plans. In the process of rehabilitation, family members support patients, accompany patients to face and cope with changes in physical, cognitive, emotional, and behavioral aspects, and help patients return to life, which is the key factor for successful rehabilitation. When family members have good coping strategies, they will also have a better mood and quality of life, which will also contribute to the rehabilitation process of patients. Therefore, it is necessary to understand the psychological coping strategies used by family caregivers in the care process and the neuropsychological function of patients. This study is divided into three stages. In the first stage, it is expected to receive 30 groups of patients and their families. Semi-structured in-depth interviews and questionnaires will be conducted for caregivers of family members with brain injury, to explore the psychological adjustment strategies developed by family caregivers in the process of care, and neuropsychological assessment will be conducted for patients to understand the impact of disease on patients' neuropsychological functions, to serve as the direction of neuropsychological intervention. In the second stage, 230 family members of patients are expected to be collected. According to the psychological adjustment strategy framework constructed in phase I, appropriate neuropsychological tests and self-report questionnaires are selected to evaluate the family members of patients, and the scale is compiled. In the third stage, it is expected to collect 60 groups of patients and their families. Through screening tests, the ecological neuropsychological intervention will be carried out for those who have an insufficient psychological function or psychological distress, and the results of neuropsychological function and psychological status before and after the intervention will be tested with evaluation tools. The objective of this study is to provide a specific framework for clinical workers and families of patients with brain injury to face difficulties together and to increase the direction of clinical psychological intervention in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patient meet ICD of brain injury
* Three months after the patient was injured
* Patient's coma score > 8
* Patient's RLAL≧5
* Patients are between 15-50 years old
* Caregiver is older than 20 years
* Caregiver can speak Mandarin or Taiwanese

Exclusion Criteria:

* Patient has developmental delay, neurological history, psychiatric history, substance abuse history, aphasia
* Caregiver has disability identification of Mental Functions and Structures of the Nervous System

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
neurophysiological indicators | 10 weeks
  EEG power in beta and theta band
neuropsychological indicators | 10 weeks
  neuropsychological test
behavioral indicators | 10 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nai-Wen, Guo, Tainan, East Dist., Taiwan

IPD SHARING:
Plan to Share IPD: Undecided